CLINICAL TRIAL: NCT06124976
Title: A Phase 2/3 Multicenter Trial Evaluating the Safety and Efficacy of ST-02 (Mucoadhesive Gemcitabine Suspension) on Ablation of Urothelial Carcinomas in the Upper Urinary Tract
Brief Title: Multicenter Clinical Trial of ST-02 for Ablation of Upper Tract Urothelial Carcinoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Peter Black, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H23-02476
Record Dates: First submitted 2023-10-27; First posted 2023-11-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Urothelial Carcinoma of the Renal Pelvis and Ureter; Transitional Cell Cancer of the Renal Pelvis and Ureter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ST-02 (Experimental): ST-02 is a new gemcitabine formulation for instillation into the upper urinary tract. Eligible participants will be enrolled and receive ST-02 once weekly for six weeks in a retrograde or antegrade fashion at the discretion of the treating urologist.
  Interventions: Drug: ST-02

INTERVENTIONS:
Drug: ST-02 — ST-02 drug instillation into the upper urinary tract (renal pelvis)

SUMMARY:
The goal of this prospective clinical trial is to investigate the safety and efficacy of ST-02 (mucoadhesive gemcitabine suspension for pyelocaliceal instillation) to treat Upper Tract Urothelial Carcinoma (UTUC) in participants who have a low-grade tumor.

The main questions this study aims to answer are:

1. Can ST-02 effectively eradicate UTUC by 3 months?
2. Is ST-02 safe for patients with UTUC?

Participants in this study will receive ST-02, a new formulation with gemcitabine once weekly for six weeks. Gemcitabine is known to be an effective drug in treating urothelial carcinoma. This new formulation will be instilled directly into the upper urinary tract (renal pelvis) and will allow the chemotherapeutic to work locally for an extended period of time. The administration process will be retrograde (via a small catheter inserted up into the kidney, under anesthesia) or antegrade (via a nephrostomy, in the clinic) once weekly for six weeks. Safety and efficacy will be monitored for up to a year after the initial response assessment.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, single-arm, open-label clinical trial assessing the safety and efficacy of ST-02 (mucoadhesive gemcitabine suspension for pyelocaliceal instillation) to chemo-ablate low-grade urothelial carcinoma of the upper urinary tract.

Participants with biopsy confirmed low-grade (LG) upper tract urothelial carcinoma (UTUC) and a tumor of 5 to 15 mm will receive 6 weekly instillations of ST-02.

The primary objective is to evaluate complete response (CR) at 3 months from the first instillation during the primary tumor evaluation (PTE) visit. This is done by ureteroscopy, and cytology, with or without biopsy if a tumor remains. If the participant presents as a CR, they will receive their first maintenance instillation of ST-02. Endoscopic monitoring of the upper tract with ureteroscopy for responders will be performed every 3 months for up to 12 months after CR, and the patient will receive a single instillation of ST-02 if no recurrence is noted each time.

Participants who do not have a CR will be treated by their physician with the standard of care, such as biopsy and laser ablation, and with any additional surgical procedure or treatment as deemed necessary by the Principal Investigator (PI).

The first stage of the trial will enroll 30 patients. If there are 8 or fewer CR among these 30 participants, the study will be stopped. Otherwise, an additional 40 participants will be accrued into phase 3, resulting in a total sample size of 70.

The durability of response, event-free survival, safety, and other outcomes will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years) male or female
* Primary or recurrent low-grade (LG), noninvasive (Ta) Upper Tract Urothelial Carcinoma (UTUC) in the renal pelvis, infundibulum, and/or calyces, based on ureteroscopy, biopsy and cytology performed within 8 weeks prior to the Screening Visit
* At least 1 measurable papillary tumor measuring 5-15 mm
* Low grade tumor(s) in the ipsilateral ureter. Every attempt should be made to ablate this tumor completely, but residual ipsilateral ureteral tumor is not an exclusion criterion.
* Prior fully ablated low grade bladder tumor(s), without the need for intravesical therapy except for single-dose chemotherapy
* A life expectancy of greater than 12 months
* No active untreated urinary tract infection (UTI) as confirmed by urine culture or urinalysis
* Women of Child bearing potential (WoCBP) and Males who have a WoCBP partner require a negative pregnancy test at the Screening visit and must use two acceptable contraceptives methods until six months post-treatment
* All sexually active males must agree to use a condom during intercourse, for at least 48 h after each instillation

Exclusion Criteria:

* Have received Bacillus Calmette - Guerin (BCG) treatment for UTUC within 6 weeks prior to Visit 1
* Pregnant (positive urine pregnancy test), planning pregnancy during trial, breast-feeding, or of childbearing potential without reliable contraception
* Unresolved infection requiring active treatment with systemic antimicrobial drugs
* History of high-grade non-muscle invasive bladder cancer within the past 6 months
* History of muscle-invasive bladder cancer during the past 2 years
* Actively being treated or intend to be treated with intravesical or systemic chemotherapy during the duration of the trial
* Urinary obstruction in the ipsilateral Upper Urinary Tract (UUT)
* Any contraindicated to gemcitabine or sensitivity to gemcitabine or any of the ST-02 ingredients
* Currently receiving another investigational agent or involved in a clinical trial with an investigational product within the past 30 days prior to Visit 1
* Active hepatitis B (chronic or acute) or active hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) rate at the Primary Tumor Evaluation (PTE) visit | 3 months
  To evaluate the tumor ablative effect (CR after 3 months) of six instillations of ST-02 in the upper urinary tract of participants with UTUC.

SECONDARY OUTCOMES:
Durable efficacy | 12 months after CR
  To evaluate the durability of tumor ablative effect 12 months after CR in participants who demonstrated complete response at 3 months after instillation of six doses of ST-02
Objective Response Rate (ORR) | 3 months
  To evaluate the objective response rate after treatment with ST-02, defined as proportion of participants with Complete Response (CR) or Partial Response (PR) at the PTE Visit
Event-Free Survival (EFS) | 15 months
  To evaluate the event-free survival after treatment with ST-02
Number of adverse event | 15 months
  To evaluate the safety and tolerability of instillation of ST-02 in participants with UTUC
Peak Plasma Concentration (Cmax) | 24 hours
  To assess the peak concentration of gemcitabine in urine and plasma at 0, 1, 2, 4 and 24 hours after instillation (10 patients, phase 2 only)
Pharmacokinetics (Tmax) | 24 hours
  To assess the time to maximal concentration of gemcitabine in urine and plasma at 0, 1, 2, 4 and 24 hours after instillation (10 patients, phase 2 only)
Rate of invasive surgery | 15 months
  To evaluate the rate of nephroureterectomy following instillation of ST-02
Clinical impact of PR in not endoscopically resectable UTUC | 3 months
  To evaluate the proportion of participants with PR whose tumors were considered not endoscopically resectable at baseline but are endoscopically resectable after treatment with ST-02

CONTACTS AND LOCATIONS:
Overall Officials: Peter Black, Dr., Principal Investigator — Vancouver Prostate Centre
Locations (4):
- Canada (4):
  - Vancouver Prostate Centre, Vancouver, British Columbia
  - Men's Health Clinic, Winnipeg, Manitoba
  - Centre of Applied Urology Research, Nova Scotia Health Authority, Halifax, Nova Scotia
  - UHN - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No